CLINICAL TRIAL: NCT02609893
Title: Pilot Treatment as Prevention for HCV Among Persons Who Actively Inject Drugs
Acronym: BYE-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Phillip Coffin, MD, MIA (Other Government)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Phillip Coffin, MD, MIA, Director, Substance Use Research Unit, San Francisco Department of Public Health
Organization: San Francisco Department of Public Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA039333 (NIH)
Record Dates: First submitted 2015-10-05; First posted 2015-11-20 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Chronic Hepatitis C
Keywords: HCV
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified Directly Observed Therapy (Active Comparator): Ledipasvir/Sofosbuvir Fixed-Dose Combination (LDV-SOF) tablet (LDV 90mg/SOF 400mg) observed daily dosing (modified for non-observed Saturday and Sunday dosing) for 8 weeks
  Interventions: Other: modified directly observed therapy (mDOT); Other: Motivational Interviewing-based counseling
- Unobserved Dosing (Active Comparator): Ledipasvir/Sofosbuvir Fixed-Dose Combination (LDV-SOF) tablet (LDV 90mg/SOF 400mg) provided weekly (7 tablets) for unobserved daily dosing for 8 weeks
  Interventions: Other: unobserved dosing; Other: Motivational Interviewing-based counseling

INTERVENTIONS:
Other: modified directly observed therapy (mDOT)
  Arms: Modified Directly Observed Therapy
Other: unobserved dosing
  Arms: Unobserved Dosing
Other: Motivational Interviewing-based counseling — Motivational Interviewing-based risk reduction and medication adherence counseling

SUMMARY:
This project is a randomized trial of two strategies to treat persons with genotype 1 HCV who currently inject drugs (PWIDs) with a once daily regime of ledipasvir-sofosbuvir (LDV-SOF) for 8 weeks. The study will enroll 30 participants and will assess the feasibility and acceptability of treating active PWIDs for HCV with LDV-SOF by modified directly observed therapy (mDOT) versus unobserved dosing, with motivational interviewing based adherence support; and assess through in-depth, semi-structured qualitative interviews, the challenges with time intensity required for mDOT and unobserved dosing interventions, and identify key factors affecting treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age;
2. 2 consecutive positive HCV RNA tests at least 6 months after estimated date of infection;
3. HCV genotype 1;
4. HCV RNA <6 million copies by Roche TaqMan Assay
5. No evidence of hepatic cirrhosis (as determined by two indices: Fib4<3.25-an accurate test for detecting cirrhosis based on age, AST, ALT and platelets [sensitivity/specificity 76-100/82-91%], confirmed by the fibrosis-cirrhosis index (FCI)<1.25 based on ALT, bilirubin, albumin and platelets [sensitivity/specificity 86/100%]);
6. Drug injection in past 30 days by self-report and physical exam evidence of injection drug use (e.g. track marks),
7. injected with others in past 12 months by self-report;
8. Lab values within acceptable range (platelets>50,000, creatinine clearance by Cockroft-Gault>30mL/min, hemoglobin >10g/dL, INR<1.5 x upper limit of normal (ULN) unless stable on anticoagulant regimen or known hemophilia, AST/ALT<10 x ULN);
9. Able to speak English;
10. No plans to leave San Francisco area for at least 9 months and either lives or works in San Francisco, or travels to San Francisco at least weekly;
11. for women of childbearing age, pregnancy test negative, not actively nursing, and agree to use birth control during treatment (although LDV-SOF has a "B" rating, consistent with no known evidence of harm, treatment is not urgent for these patients so we will err on the side of caution).

Exclusion Criteria:

1. HIV+ by rapid test or pooled viral load;
2. HBV surface antigen +;
3. Non-definitive HCV genotype results;
4. Previously received treatment for HCV (interferon, ribavirin, or DAA);
5. Taking medications that affect pharmacokinetics of LDV-SOF (proton-pump inhibitors, anticonvulsants [phenobarbital, phenytoin, carbamazepine, oxcarbazepine], rifamycins, rosuvastatin, herbs [St. John's wort, silymarin, echinacea]);
6. History of any of the following:

   1. Current gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug
   2. History of hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage)
   3. History of solid organ or bone marrow transplantation.
   4. Current treatment for cancer
7. Chronic liver disease for non HCV reason, except iron overload (e.g., Wilson's disease, alfa 1 antitrypsin deficiency, cholangitis);
8. Use of any prohibited concomitant medications as described in Section 5.2 within 21 days of the Day 1 visit; and
9. Known hypersensitivity to LDV, SOF, the metabolites, or formulation excipients.
10. No other conditions that preclude study involvement as determined by PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-12; Primary Completion 2018-04 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Number of people who inject drugs (PWIDs) with HCV who were recruited and retained | 44 weeks
  To determine the feasibility of treating active PWIDs for HCV with LDV-SOF by mDOT versus unobserved dosing based on proportion eligible and enrolled among those screened and completion rates overall and by arm.
Medication adherence to study drug | 44 weeks
  To evaluate the acceptability of mDOT versus unobserved dosing, the percent of treatment medication adherence to LDV-SOF, as measured by the percent of doses taken overall (observed and unobserved), will be assessed using DOT doses and weekend Wise Pill data for the mDOT arm, and WisePill data for the unobserved dosing arm.
Challenges of medication adherence | 44 weeks
  To assess through in-depth, semi-structured qualitative interviews, the challenges with time intensity required for mDOT versus unobserved dosing for PWIDs treated with LDV-SOF.

SECONDARY OUTCOMES:
SVR (end-of-treatment response) | 12 weeks
  We will compare the proportion of participants with undetectable HCV RNA at week 8 and post-treatment week 12 between arms.
SOF/metabolite levels | 8 weeks
  SOF/metabolite-positivity rates will be calculated by week in both arms.
HCV relapse and reinfection | 36 weeks
  Among participants who achieve SVR, we will determine the proportion who experience HCV relapse and reinfection at post-treatment week 36, overall and by arm.
Social and injector networks of participants | 44 weeks
  We will characterize injector network sizes at baseline and follow-up through ACASI surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip O Coffin, M.D., Principal Investigator — San Francisco Department of Public Health; Emily Behar, MS, Study Director — San Francisco Department of Public Health
Locations (1):
- Substance Use Research Unit, San Francisco, California, United States

REFERENCES:
- [Derived] Coffin PO, Santos GM, Behar E, Hern J, Walker J, Matheson T, Kinnard EN, Silvis J, Vittinghoff E, Fox R, Page K. Randomized feasibility trial of directly observed versus unobserved hepatitis C treatment with ledipasvir-sofosbuvir among people who inject drugs. PLoS One. 2019 Jun 3;14(6):e0217471. doi: 10.1371/journal.pone.0217471. eCollection 2019. PMID 31158245